CLINICAL TRIAL: NCT06000020
Title: Leave or Laparoscopic Appendectomy With Normal Findings - a Regional Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Nordsjaellands Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LapApp
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Appendicitis Acute
Keywords: Laparoscopic appendectomy; Normal findings
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic laparoscopy: Diagnostic laparoscopy on suspicion of acute appendicitis with normal intraoperative findings (including mesenteric adenitis).
- Laparoscopic appendectomy: Laparoscopic appendectomy despite normal intraoperative findings (including mesenteric adenitis) and histopathology showing a normal appendix.
  Interventions: Procedure: Laparoscopic appendectomy

INTERVENTIONS:
Procedure: Laparoscopic appendectomy — Laparoscopic appendectomy as performed as standard world wide. Division of the appendix with laparoscopic stapler.
  Groups: Laparoscopic appendectomy

SUMMARY:
Based on a regional cohort, this study we will try to demonstrate the superiority of routine laparoscopic appendectomy vs. leaving an intraoperative assessed normal appendix in situ in cases of normal findings at diagnostic laparoscopy. If routine laparoscopic appendectomy is not superior, we will recommend leaving the "normal" appendix in situ.

DETAILED DESCRIPTION:
The study is a retrospective cohort study with a superiority design. It will be carried out at the surgical departments of the four public university hospitals providing emergency surgical service to the entire population of 1,8 million in the Capital Region of Denmark.

On March 17, 2017, a new electronic health record (EHR) had been implemented at three of the hospital, while it was implemented at Copenhagen University Hospital - Bispebjerg on May 20, 2017. These dates mark the start of the inclusion period for each hospital, while the inclusion period ended April 1, 2021 for all four hospitals.

The "snap boards" covering the relevant operation rooms at the four hospitals will be systematically review. For all cases, where diagnostic laparoscopy was performed on suspicion of acute appendicitis, the EHR will be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic laparoscopy with normal intraoperative findings (including mesenteric adenitis
* Laparoscopic appendectomy and a histopathological normal appendix and otherwise normal intraoperative findings (including mesenteric adenitis)

Exclusion Criteria:

* Diagnostic laparoscopy with abnormal intraoperative findings.
* Laparoscopic appendectomy and a histopathological non-normal appendix.
* Laparoscopic appendectomy and a histopathological normal appendix and abnormal intraoperative findings.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing diagnostic laparoscopy on suspicion of acute appendicitis
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Risk of surgery on suspicion of acute appendicitis | 3 years
  Laparoscopy or laparotomy after surgery on suspicion of acute appendicitis
Risk of surgery on suspicion of acute appendicitis | 5 years
  Laparoscopy or laparotomy after surgery on suspicion of acute appendicitis

SECONDARY OUTCOMES:
Reintervention | 30 days
  Laparoscopy or laparotomy due to complications
Postoperative complications | 30 days
  Postoperative complications according to the 'Clavien-Dindo classification'
Length of stay | 30 days
  Time from index surgery to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, Ph.D., Study Chair — cabertelsen@gmail.com
Locations (4):
- Denmark (4):
  - Copenhagen University Hospital - Bispebjerg, Copenhagen NV
  - Copenhagen University Hospital - Herlev, Herlev
  - Copenhagen University Hospital - North Zealand, Hillerød
  - Copenhagen University Hospital - Hvidovre, Hvidovre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaunoo SS, Hale AL, Masters JP, Jaunoo SR. An international survey of opinion regarding investigation of possible appendicitis and laparoscopic management of a macroscopically normal appendix. Ann R Coll Surg Engl. 2012 Oct;94(7):476-80. doi: 10.1308/003588412X13373405385377. PMID 23031764
- [Background] Di Saverio S, Birindelli A, Kelly MD, Catena F, Weber DG, Sartelli M, Sugrue M, De Moya M, Gomes CA, Bhangu A, Agresta F, Moore EE, Soreide K, Griffiths E, De Castro S, Kashuk J, Kluger Y, Leppaniemi A, Ansaloni L, Andersson M, Coccolini F, Coimbra R, Gurusamy KS, Campanile FC, Biffl W, Chiara O, Moore F, Peitzman AB, Fraga GP, Costa D, Maier RV, Rizoli S, Balogh ZJ, Bendinelli C, Cirocchi R, Tonini V, Piccinini A, Tugnoli G, Jovine E, Persiani R, Biondi A, Scalea T, Stahel P, Ivatury R, Velmahos G, Andersson R. WSES Jerusalem guidelines for diagnosis and treatment of acute appendicitis. World J Emerg Surg. 2016 Jul 18;11:34. doi: 10.1186/s13017-016-0090-5. eCollection 2016. PMID 27437029
- [Background] Bakker OJ, Go PM, Puylaert JB, Kazemier G, Heij HA; Werkgroep richtlijn Diagnostiek en behandeling van acute appendicitis. [Guideline on diagnosis and treatment of acute appendicitis: imaging prior to appendectomy is recommended]. Ned Tijdschr Geneeskd. 2010;154:A303. Dutch. PMID 21262032
- [Background] Lee M, Paavana T, Mazari F, Wilson TR. The morbidity of negative appendicectomy. Ann R Coll Surg Engl. 2014 Oct;96(7):517-20. doi: 10.1308/003588414X13946184903801. PMID 25245730
- [Background] Bijnen CL, Van Den Broek WT, Bijnen AB, De Ruiter P, Gouma DJ. Implications of removing a normal appendix. Dig Surg. 2003;20(2):115-21. doi: 10.1159/000069386. PMID 12686778
- [Background] Gough IR, Morris MI, Pertnikovs EI, Murray MR, Smith MB, Bestmann MS. Consequences of removal of a "normal" appendix. Med J Aust. 1983 Apr 16;1(8):370-2. doi: 10.5694/j.1326-5377.1983.tb99414.x. PMID 6835144
- [Background] Sorensen AK, Bang-Nielsen A, Levic-Souzani K, Pommergaard HC, Jorgensen AB, Tolstrup MB, Rud B, Kovacevic B, Bulut O. Readmission and reoperation rates following negative diagnostic laparoscopy for clinically suspected appendicitis: The "normal" appendix should not be removed - A retrospective cohort study. Int J Surg. 2019 Apr;64:1-4. doi: 10.1016/j.ijsu.2019.02.001. Epub 2019 Feb 12. PMID 30769215